CLINICAL TRIAL: NCT04996524
Title: Epidural vs. Systemic Analgesia in the Intensive Care Unit: Retrospective Study
Brief Title: Epidural vs. Systemic Analgesia in the Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0158-21-MMC
Record Dates: First submitted 2021-07-29; First posted 2021-08-09 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Patients With Acute Pain Admitted to the Intensive Care Unit
Keywords: acute pain, epidural analgesia, intensive care unit
MeSH Terms: conditions — Acute Pain | interventions — Analgesia, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- epidural analgesia group (Experimental)
  Interventions: Drug: epidural analgesia
- systemic analgesia group (No Intervention)

INTERVENTIONS:
Drug: epidural analgesia — Patients recieving epidural analgesia instead of systemic analgesia for acute pain in the intensive care unit
  Arms: epidural analgesia group

SUMMARY:
Many patients admitted to the general intensive care unit suffer from pain, whether acute or chronic. Those patients include post-operative patients, multi trauma, acute pancreatitis and patients with multiple rib fractures. Most patients in the intensive care unit, whether intubated and ventilated or not, are treated with systemic analgesic drugs, usually given intravenously, enterally, or trans dermally (fentanyl patches).

Continuous epidural anesthesia has been shown in several studies to have an advantage over systemic analgesia in specific conditions, such as pancreatitis, multiple rib fractures and upper abdominal surgeries. Some of its benefits include improved gastrointestinal motility (reduction of ileus rates), decreased thromboembolic events (DVT) and better quality of pain control. In intubated and ventilated patients, continuous epidural anesthesia may reduce the amount of required systemic sedation. Reducing the amount of sedation may contribute to a decrease in delirium rates, shortening the time to extubation and reducing other adverse effects associated with high requirements of sedation drugs (such as a decrease in blood pressure).

Most of the studies comparing systemic analgesia to epidural analgesia examined a population of patients hospitalized in the surgical ward, post breast, abdominal or orthopedic surgeries of the pelvis and lower extremities, or due to other conditions such as pancreatitis or multiple rib fractures. There are almost no studies that have examined the effectiveness of epidural analgesia in patients admitted to the intensive care unit, including sedated and ventilated patients, compared with systemic analgesia.

From 2011 until today, our intensive care unit has admitted about 300 patients who were treated with continuous epidural analgesia. In this study we would like to compare them to another group of patients (about 300 patients as well), who were admitted to the unit for similar etiologies (post-operative, multi- trauma, pancreatitis, etc.), and to observe differences between the groups. We would like to examine differences in mortality within 28 days, as well as differences in morbidity, such as the level of analgesia and delirium rates between groups.

ELIGIBILITY:
Inclusion Criteria:Patients aged 18-99, admitted to the General Intensive Care Unit from January 2011 to June 2021 (inclusive), due to a medical condition that may expose them to significant pain during hospitalization: chest, abdominal, pelvic or lower extremity surgery, pancreatitis, multiple rib fractures, trauma including chest, abdominal, pelvic, or lower limb trauma, and treated with epidural or systemic anesthesia during their stay in the unit.

-

Exclusion Criteria:Patients not admitted for the above reasons. -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 647 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
delirium score | 6 months post ICU admission
  To compare delirium score, as measured by RASS score, between the epidural group and the systemic analgesia group

SECONDARY OUTCOMES:
pain score | 6 months post ICU admission
  To compare pain score, as measured by VAS score, between the epidural group and the systemic analgesia group

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center Kfar Saba, Kfar Saba, Israel